CLINICAL TRIAL: NCT03022149
Title: Remote Ischemic Preconditioning for Subcortical Vascular Dementia
Acronym: RIPSVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Junwei Hao, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2016-YX-042
Record Dates: First submitted 2016-12-30; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Subcortical Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doctormate® (200mmHg) (Experimental): Patients will be treated with Renqiao Remote Ischemic Conditioning Device (Doctormate®) (200mmHg) once daily for 6 months
  Interventions: Device: Doctormate® (200mmHg)
- Doctormate® (60mmHg) (Sham Comparator): Patients will be treated with Renqiao Remote Ischemic Conditioning Device (Doctormate®) (60mmHg) once daily for 6 months
  Interventions: Device: Doctormate® (60mmHg)

INTERVENTIONS:
Device: Doctormate® (200mmHg) — Limb ischemia was induced by Renqiao Remote Ischemic Conditioning Device (Doctormate®) inflating tourniquets to 200mmHg.
  Arms: Doctormate® (200mmHg)
Device: Doctormate® (60mmHg) — Limb ischemia was induced by Renqiao Remote Ischemic Conditioning Device (Doctormate®) inflating tourniquets to 60mmHg.
  Arms: Doctormate® (60mmHg)

SUMMARY:
The purpose of this study is to determine whether the remote ischemic preconditioning are effective in the treatment of mild to moderate vascular dementia.

DETAILED DESCRIPTION:
In this randomized, double-blind, placebo-controlled trial, the investigators enrolled 52 participants aged 50-80 years. The participants had a diagnosis of subcortical vascular dementia at the neurology department of Tianjin medical university general hospital. Inclusion criteria included a clinical dementia rating 1-2; a mini-mental state examination score 15-26; and brain magnetic resonance imaging consistent with subcortical ischemic small vessel disease. All participants received standard medical management.Participants in the remote ischemic preconditioning group underwent 5 brief cycles consisting of bilateral upper limb ischemia followed by reperfusion. The remote ischemic precondition procedure was performed once daily over 180 consecutive days. Cognitive impairment assessment scale ( Hopkins Verbal Learning Test,HVLT;Symbol digital modalities tes,SDMT;judgement line orientation, JLO;trail making test A and B,TMT-A/B;chinese word fluency test;Activity of Daily Living Scale,ADL;Neuropsychiatric Inventory,NPI), serological inflammatory markers:hypersensitive C-reactive protein（hs-CRP）、plasma tumor necrosis factor-α(TNF-α)、interleukin-1β(IL-1β)、interleukin-6 (IL-6)、α1-antichymotrypsin),and MRI diffusion tensor imaging, DTI were compared with the untreated control group.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of vascular dementia
2. In three months without cerebral infarction
3. MMSE 15 to 26 points;CDR 1-2 points;MoCA < 26 points
4. MRI showed subcortical ischemic cerebrovascular disease.

Exclusion Criteria:

1. AD 、 FTD, DLB and other causes of dementia.
2. Cortical/subcortical infarction
3. Cortex watershed infarction
4. Cerebral hemorrhage
5. Hydrocephalus
6. Other special causes of white matter lesions such as multiple sclerosis, sarcoidosis, radiation encephalopathy, etc.
7. Cannot complete aphasia neuropsychological assessment.
8. Genetic or inflammatory small vascular disease.
9. Serious cardiovascular, lung, liver, kidney, endocrine, such as infection disease.
10. Alcohol poisoning;
11. Cancer
12. Hypothyroidism
13. Schizophrenia;Hamilton depression rating scale > 17 points.
14. Can not complete MRI.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment assessment scale-HVLT | At the first day/sixth month after randomization
  Comparing two groups of participants score changes in Short-term auditory verbal memory、learning rate and learning strategies.
Cognitive impairment assessment scale-SDMT | At the first day/sixth month after randomization
  Comparing two groups of participants score changes in-attention.
Cognitive impairment assessment scale-JLO | At the first day/sixth month after randomization
  Comparing two groups of participants score changes in spatial perception and orientation ability.
Cognitive impairment assessment scale-ADL | At the first day/sixth month after randomization
  Comparing two groups of participants score changes in daily life ability.
Cognitive impairment assessment scale-TMT | At the first day/sixth month after randomization
  Comparing two groups of participants score changes in this test.This test reflects notice, order, mental flexibility, visual search and motor function, and set transfer (set shifting), at the same time reflect the hand-eye coordination, spatial perception and pay attention to ability.
Cognitive impairment assessment scale-NPI | At the first day/sixth month after randomization
  Comparing two groups of participants score changes in mental behavior symptoms.
Cognitive impairment assessment scale-Chinese auditory learning test | At the first day/sixth month after randomization
  Comparing two groups of participants score changes in speech ACTS and breadth of knowledge.

SECONDARY OUTCOMES:
Serological inflammatory markers-hs-CRP | At the fist day/sixth month after randomization
  Collecte venous blood from two groups of paticipants at the first day/sixth month,detect the inflammatory factors by ELISA and compare the changes between the two groups.
Serological inflammatory markers-TNF-a | At the fist day/sixth month after randomization
  Collecte venous blood from two groups of paticipants at the first day/sixth month,detect the inflammatory factors by ELISA and compare the changes between the two groups.
Serological inflammatory markers-IL - 1b | At the fist day/sixth month after randomization
  Collecte venous blood from two groups of paticipants at the first day/sixth month,detect the inflammatory factors by ELISA and compare the changes between the two groups.
Serological inflammatory markers-IL - 6 | At the fist day/sixth month after randomization
  Collecte venous blood from two groups of paticipants at the first day/sixth month,detect the inflammatory factors by ELISA and compare the changes between the two groups.
Serological inflammatory markers-ACT | At the fist day/sixth month after randomization
  Collecte venous blood from two groups of paticipants at the first day/sixth month,detect the inflammatory factors by ELISA and compare the changes between the two groups.
Imaging markers-DTI | At the fist day/sixth month after randomization
  To evaluate two groups of whole brain white matter (whole brain white matter, WBWM) and apparent normal white matter (normal appearing white matter, NAWM) difference of MD and FA before and after the treatment , to evaluate whether the treatment group more helpful to improve the neural axon damage.
Imaging markers-Routine MRI | At the fist day/sixth month after randomization
  To evaluate two sets of T2 weighted white matter lesions volume (T2 weighted lesion volume, T2WLV) before and after the treatment.

OTHER OUTCOMES:
Laboratory examination of the urine routine | At the first month/third month after randomization
Laboratory examination of the blood routine | At the first month/third month after randomization
Laboratory examination of the blood coagulation function | At the first month/third month after randomization
Laboratory examination of the liver function | At the first month/third month after randomization
Laboratory examination of the kidney function | At the first month/third month after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, PHD, MD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liao Z, Bu Y, Li M, Han R, Zhang N, Hao J, Jiang W. Remote ischemic conditioning improves cognition in patients with subcortical ischemic vascular dementia. BMC Neurol. 2019 Aug 23;19(1):206. doi: 10.1186/s12883-019-1435-y. PMID 31443692